CLINICAL TRIAL: NCT06013163
Title: Control Of BioEquivalence With Xenical (COBEX): A Phase I, Randomised, Active-control Study to Evaluate EMP22 Pharmacodynamics and EMP16 Pharmacokinetics Versus Xenical® in Healthy Volunteers
Brief Title: A Phase 1 Study to Evaluate EMP22 PD and EMP16 PK Versus Xenical® in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Empros Pharma AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: EP-004; 2023-505671-74-00 (Other: EU Trial no)
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Overweight or Obesity
Keywords: Overweight, Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: In Part I (single-blind), EMP22 (120 mg orlistat) and orlistat in its conventional form (Xenical®, 120 mg orlistat) will be taken 3 times daily (ter in die [TID]) together with the 3 main daily meals for two 9-day treatment periods in a cross-over manner.
  In Part II (open-label), single doses of EMP16 (120 mg orlistat/40 mg acarbose) and Xenical® (120 mg orlistat) will be taken together with breakfast on 2 separate days.
Who Masked: Participant
Masking Description: Part I: EMP22 and Xenical® have different strengths of orlistat, 60 mg and 120 mg, respectively. In order to maintain the blind, the IMP will be administered as follows:
  * EMP22 60 mg orlistat, 2 capsules TID.
  * Xenical® 120 mg orlistat 1 capsule + placebo 1 capsule TID. EMP22, Xenical® and placebo will be identical in appearance.
  Part II will be open-label, i.e., the Investigator, trial staff and trial participants will know which treatment, EMP16 or Xenical®, that is given at each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Xenical - EMP22 part 1 crossover blinded (Active Comparator): After a 5-day diet run-in period, orlistat in its conventional form (Xenical®, 120 mg orlistat) will be taken 3 times daily (ter in die [TID]) together with the 3 main daily meals for a 9-day treatment period. After a 4-to-14-day wash-out period; EMP22 (120 mg modified release orlistat) will be taken TID together with the 3 main daily meals for a 9-day treatment period.
  Interventions: Drug: Xenical® vs EMP 22
- EMP22 - Xenical part 1 crossover blinded (Active Comparator): After a 5-day diet run-in period, EMP22 (120 mg modified release orlistat) will be taken 3 times daily (ter in die [TID]) together with the 3 main daily meals for a 9-day treatment period. After a 4-to-14-day wash-out period; orlistat in its conventional form (Xenical®, 120 mg orlistat) will be taken TID together with the 3 main daily meals for a 9-day treatment period.
  Interventions: Drug: EMP 22 vs Xenical®
- EMP16 - Xenical part 2 sequential open label (Active Comparator): Single dose of EMP16 (120 mg orlistat/40 mg acarbose) will be taken together with breakfast during one PK study day. After a 4-to-14-day wash-out period, Xenical® (120 mg orlistat) will be taken together with breakfast during one PK study day.
  Interventions: Drug: EMP 16 vs Xenical®

INTERVENTIONS:
Drug: Xenical® vs EMP 22 — Each participant will first use Xenical® TID for 9 days and then EMP22TID for 9 days (in total 27 doses of each drug).
  Other Names: Part I
  Arms: Xenical - EMP22 part 1 crossover blinded
Drug: EMP 22 vs Xenical® — Each participant will first use EMP22 TID for 9 days and then Xenical® TID for 9 days (in total 27 doses of each drug).
  Other Names: Part I
  Arms: EMP22 - Xenical part 1 crossover blinded
Drug: EMP 16 vs Xenical® — Each participant will receive a single dose of EMP16 and then a single dose of Xenical®.
  Other Names: Part II
  Arms: EMP16 - Xenical part 2 sequential open label

SUMMARY:
This Phase I, active-controlled, randomised trial will be conducted in 2 parts. Part I aims to confirm the PD equivalence of EMP22 and Xenical® based on percent fecal fat excretion at steady state. EMP22 (also referred to as MR orlistat) has the same MR properties as EMP16 but lacks the acarbose component. Part II will explore the PK properties of EMP16 alone and vs. Xenical®. Part I will be conducted in a single-blind, cross-over fashion while Part II will have an open-label, fixed-sequence design. Healthy volunteers will be recruited to the trial.

DETAILED DESCRIPTION:
Approximately 35 participants are planned to be screened to achieve 20 randomised participants and at least 16 evaluable participants in Part I.

All participants who complete Part I will continue in Part II.

Each participant is expected to participate in the trial for approximately 9 to 13 weeks (depending on the length of each wash-out period), including a 28-day screening period.

Part I: Participants will self-administer EMP22 for 9 days and Xenical® for 9 days (TID dosing) at home. EMP22 and Xenical® should be taken halfway through each of the 3 main meals during the day (breakfast, lunch, dinner) with approximately 50 to 200 mL water.

EMP22 and Xenical® have different strengths of orlistat, 60 mg and 120 mg, respectively. In order to maintain the blind for the participants, the IMP will be administered as follows:

* EMP22 60 mg orlistat, 2 capsules TID.
* Xenical® 120 mg orlistat 1 capsule + placebo 1 capsule TID.

Part II: Following an overnight fast of at least 8 hours and a light standardised breakfast upon admission (approximately 2 hours prior to dose), EMP16 will be taken halfway through a regular standardised breakfast (5 minutes after the start of the meal, which is expected to be finished in 10 minutes) with approximately 50 to 200 mL water. After a 4-14 day washout, the same procedure will be repeated using Xenical® .

The participants will receive a single dose dose of EMP16 (2 capsules, each of 60 mg) and a single dose of Xenical® (1 capsule, 120 mg).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the trial.
2. Healthy male or female aged 20 to 55 years inclusive.
3. Participants with a BMI between 20 and 27 kg/m² or participants with a BMI >27 kg/m2 and normal body fat composition (10 to 25% for men and 20 to 30% for women measured using a bioimpedance scale) at screening.
4. Weight stable (<5% self-reported change during the previous 3 months preceding screening).
5. Participants with a self-perceived normality in defecation habits, normally with a stool frequency of at least once daily.
6. Medically healthy participant without abnormal clinically significant medical history, physical findings, vital signs, electrocardiogram (ECG) and laboratory values at the time of the screening visit, as judged by the Investigator.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or influence the results or the participant's ability to participate in the trial including but not limited to:

   * GI problems/diseases, e.g. inflammatory bowel diseases and irritable bowel syndrome (IBS).
   * Cholestasis.
   * Previous GI surgery that might influence GI function significantly, such as previous bariatric surgery, and previous gallbladder surgery as judged by the investigator.
   * Vitamin B12 deficiency or other signs of achlorhydria.
   * Chronical malabsorption syndrome.
   * History of severe allergic, cardiac or hepatic disease.
2. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
3. Malignancy within the past 5 years, with the exception of in situ removal of basal cell carcinoma.
4. Any planned major surgery within the duration of the trial.
5. Participants who are pregnant, currently breastfeeding, or intend to become pregnant during the course of the trial.
6. Any positive result at the screening visit for serum hepatitis B surface antigen, hepatitis C antibodies and/or human immunodeficiency virus (HIV).
7. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG at the screening visit, as judged by the Investigator.
8. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to drugs with a similar chemical structure or class as orlistat or acarbose.
9. Regular use of any prescribed or non-prescribed medications (including, but not limited to, antacids, analgesics, herbal remedies, vitamins and minerals) within 2 weeks prior to the first administration of IMP except as outlined in Section 9.6.2.3.
10. Administration of another new chemical entity (defined as a compound which has not been approved for marketing) or has participated in any other clinical trial that included drug treatment within 3 months of the first administration of IMP in this trial. Subjects consented and screened but not dosed in previous studies are not excluded.
11. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than 3 times/week is allowed before the screening visit.
12. Positive screening result for drugs of abuse or alcohol at the screening visit.
13. History of alcohol abuse or excessive intake of alcohol, as judged by the Investigator.
14. Presence or history of drug abuse, as judged by the Investigator.
15. History of, or current use of anabolic steroids, as judged by the Investigator.
16. Excessive caffeine consumption defined by a daily intake of > 5 cups (1 cup = approximately 240 mL) of caffeine containing beverages, as judged by the Investigator.
17. Plasma donation within 1 month of screening or blood donation (or corresponding blood loss) during the last 3 months prior to screening.
18. The Investigator considers the participant unlikely to comply with trial procedures, restrictions and requirements.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The percent of faecal fat | Day -2 , Day -1 , and between the morning of Day 9 and Day 10.
  The percent of faecal fat excretion expressed as a ratio of the amount of fat excretion over a 24-hour period at steady-state relative to the amount of daily ingested fat.

SECONDARY OUTCOMES:
Cmax - to explore the PK properties of EMP16 | 12 hour for each day of treatment
  Cmax for orlistat and acarbose
Tmax - to explore the PK properties of EMP16 | 12 hour for each day of treatment
  Tmax for orlistat and acarbose
AUC0-t - to explore the PK properties of EMP16 | 12 hour for each day of treatment
  AUC0-t for orlistat and acarbose
Cmax - to compare the bioavailability of orlistat in EMP16 and Xenical® | 12 hour for each day of treatment
  Cmax for orlistat
Tmax - to compare the bioavailability of orlistat in EMP16 and Xenical® | 12 hour for each day of treatment
  Tmax for orlistat
AUC0-t - to compare the bioavailability of orlistat in EMP16 and Xenical® | 12 hour for each day of treatment
  AUC0-t for orlistat

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Holmbäck, Study Chair — Empros Pharma
Locations (1):
- CTC Clinical Trial Consultanta AB, Uppsala, Sweden